CLINICAL TRIAL: NCT02192164
Title: Non-interventional Study Of The Effect Of Smoking Status Of The Patient On The Success Of Etanercept Therapy In Psoriasis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801365
Record Dates: First submitted 2014-04-11; First posted 2014-07-16 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-04

CONDITIONS: Plaque Psoriasis
Keywords: plaque psoriasis; smoking; etanercept
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: smoking questionnaire — patients fill in a smoking questionnaire about their smoking habits

SUMMARY:
Pilot observational study to describe the relationship between the smoking status of a psoriatic individual and the success of etanercept therapy in psoriasis treatment

DETAILED DESCRIPTION:
non-interventional study There is no sampling

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of chronic plaque type psoriasis for at least 6 months as determined by the subjects medical history, and confirmation of the diagnosis through physical examination by the investigator Patients who are scheduled by their dermatologist to initiate treatment with Etanercept

Exclusion Criteria:

Previous or current treatment with antipsoriatic biologic drugs, such as etanercept, infliximab, adalimumab, ustekinumab, alefacept, efalizumab Chronic or acute infections requiring intravenous or oral anti-infectives within 14 days prior to the Baseline visit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: etanercept treated plaque psoriasis patients
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Hungary (8):
  - Semmelweis University, Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum/Bor- es Nemikortani Klinika, Debrecen
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Bacs-Kiskun Megyei Onkormanyzat Korhaza Szegedi Tudomanyegyetem AOK Oktato Korhaza, Kecskemét
  - Semmelweis Korhaz-Rendelointezet, Miskolc
  - Pecsi Tudomanyegyetem, Br-, Nemikortani es Onkodermatologiai Klinika, Pécs
  - Medical University of Szeged, Szeged
  - Vas Megyei Markusovszky Korhaz/Borgyogyaszati Osztaly, Szombathely

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801365&StudyName=Non-interventional%20Study%20of%20the%20Effect%20of%20Smoking%20Status%20of%20the%20Patient%20on%20the%20Success%20of%20Etanercept%20Therapy%20in%20Psoriasis%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Participants who had moderate to severe plaque psoriasis and commenced treatment based on treating physician's discretion as per Summary of Product Characteristics (SmPC) were observed prospectively for 24 weeks. According to SmPC, recommended dose included etanercept 25 milligram (mg) twice weekly, 50 mg once weekly or 50 mg twice weekly subcutaneous injection.
Period: Overall Study
Arm/Group | Etanercept
Started | 126
Etanercept Treated Population | 112
Completed | 112
Not Completed | 14
Not completed — Other | 8
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 4
Not completed — Did not meet the exclusion criteria | 1

BASELINE CHARACTERISTICS:
Population: All treated participants with available post-baseline documentation.
Arm/Group | Etanercept
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.37 (15.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 67

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Psoriasis Assessment and Severity Index (PASI) Score at Week 24
Description: PASI score is the combined assessment of lesion severity and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u], trunk [t], legs [l]); each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated: 0 (no involvement) to 6 (90-100 percent involvement), severity estimated by clinical signs: erythema (E), induration (I), scaling (S); 5 point scale: 0 (no involvement) to 4 (very marked involvement). Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4.
Time Frame: Baseline (Day 1), Week 24
Population: All treated participants with available post-baseline documentation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Etanercept: Non Smokers: Participants who had never smoked and those who had quitted smoking at least 1 year prior to the study and had moderate to severe plaque psoriasis, commenced treatment based on treating physician's discretion as per SmPC were observed prospectively for 24 weeks. According to SmPC, recommended dose included etanercept 25 mg twice weekly, 50 mg once weekly or 50 mg twice weekly subcutaneous injection.
- Etanercept: Smokers: Participants who were smokers during the study and had moderate to severe plaque psoriasis, commenced treatment based on treating physician's discretion as per SmPC were observed prospectively for 24 weeks. According to SmPC, recommended dose included etanercept 25 mg twice weekly, 50 mg once weekly or 50 mg twice weekly subcutaneous injection.
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Number analyzed (Participants) | 86 | 26
units on a scale
  Baseline | 21.02093 (6.298742) | 20.40769 (4.991266)
  Change at Week 24 | -18.40349 (6.606279) | -15.64615 (8.649496)
Statistical Analysis 1: Comparison: Etanercept: Non Smokers vs Etanercept: Smokers; Test type: Superiority or Other; Mean Difference (Net) = -2.757334, 95% CI 2-sided [-5.916307 to 0.401638], Standard Error of Mean 1.594019

2. Secondary Outcome: Change From Baseline in Psoriasis Assessment and Severity Index (PASI) Score at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: All treated participants with available post-baseline documentation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Number analyzed (Participants) | 86 | 26
units on a scale | -18.18837 (6.236787) | -17.27692 (6.819402)
Statistical Analysis 1: Comparison: Etanercept: Non Smokers vs Etanercept: Smokers; Test type: Superiority or Other; Mean Difference (Net) = -0.911449, 95% CI 2-sided [-3.73847 to 1.915572], Standard Error of Mean 1.426517

3. Secondary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 75 (PASI75) Response at Week 12 and 24
Description: PASI score is the combined assessment of lesion severity and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u], trunk [t], legs [l]); each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated: 0 (no involvement) to 6 (90-100 percent involvement), severity estimated by clinical signs: erythema (E), induration (I), scaling (S); 5 point scale: 0 (no involvement) to 4 (very marked involvement). Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4. PASI75 response was defined as at least a 75 percent (%) reduction in PASI relative to Baseline.
Time Frame: Week 12, 24
Population: All treated participants with available post-baseline documentation.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Number analyzed (Participants) | 86 | 26
percentage of participants
  Week 12 | 82.56 (6.937556) | 76.92 (8.768914)
  Week 24 | 86.05 | 69.23

4. Secondary Outcome: Percent Change From Baseline in Psoriasis Assessment and Severity Index (PASI) at Week 12 and 24
Description: Percentage improvement in PASI score from baseline was calculated at Week 12 and 24 in terms of percent change from baseline. PASI score is the combined assessment of lesion severity and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u], trunk [t], legs [l]); each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated: 0 (no involvement) to 6 (90-100 percent involvement), severity estimated by clinical signs: erythema (E), induration (I), scaling (S); 5 point scale: 0 (no involvement) to 4 (very marked involvement). Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4.
Time Frame: Baseline, Week 12, 24
Population: All treated participants with available post-baseline documentation.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Number analyzed (Participants) | 86 | 26
percent change
  Week 12 | 0.139 (0.163) | 0.168 (0.218)
  Week 24 | 0.120 (0.196) | 0.257 (0.358)

5. Other Pre Specified Outcome: Smoking Habit Questionnaire: Smoking Status of Participants
Description: Smoking habit questionnaire that was conducted on Day 1, assessed the data on smoking status of participants. Smoking status of participants was classified as never smoked, current smokers, and former smokers. Former smokers were defined as those participants who had stopped smoking at least 1 year prior to the study.
Time Frame: Day 1
Population: All treated participants with available post-baseline documentation.
Measure: Number; unit: participants
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Number analyzed (Participants) | 86 | 26
participants
  Never smoke | 51 | 0
  Current smokers | 0 | 26
  Former smokers | 35 | 0

6. Other Pre Specified Outcome: Smoking Habit Questionnaire: Mean Age of Participants at Which Cigarette Smoking Started and Quitted
Description: Smoking habit questionnaire that was conducted on Day 1, assessed the data on smoking which included the age of participants at which they started smoking and the age at which they quitted smoking. Former smokers were defined as those participants who had stopped smoking at least 1 year prior to the study.
Time Frame: Day 1
Population: All treated participants with available post-baseline documentation. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for each arm. Data for this outcome measure was planned to be analyzed in smokers and former smokers.
Measure: Mean (Standard Error); unit: years
Groups:
- Etanercept: Former Smoker + Smoker: Participants who were smokers during the study and those who had quitted smoking at least 1 year prior to the study and had moderate to severe plaque psoriasis, commenced treatment based on treating physician's discretion as per SmPC were observed prospectively for 24 weeks. According to SmPC, recommended dose included etanercept 25 mg twice weekly, 50 mg once weekly or 50 mg twice weekly subcutaneous injection.
Arm/Group | Etanercept: Former Smoker + Smoker
Number analyzed (Participants) | 61
years
  Age when participants started smoking (n =61) | 18.55738 (0.7493256)
  Age when participants quitted smoking (n =35) | 21.25714 (2.165948)

7. Other Pre Specified Outcome: Smoking Habit Questionnaire: Mean Duration of Smoking Among Participants
Description: Smoking habit questionnaire which was conducted on Day 1, assessed the data on smoking which included the mean duration (in years) of smoking among participants. Former smokers were defined as those participants who had stopped smoking at least 1 year prior to the study.
Time Frame: Day 1
Population: All treated participants with available post-baseline documentation. Here, 'N' signifies those participants who were evaluable for this measure. Data for this outcome measure was planned to be analyzed in smokers and former smokers.
Measure: Mean (Standard Error); unit: years
Arm/Group | Etanercept: Former Smoker + Smoker
Number analyzed (Participants) | 61
years | 21 (1.604808)

ADVERSE EVENTS:
Description: Due to non-interventional nature of the study, safety data was not planned to be collected.
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Prioritization of outcome measures as primary and secondary was based on the study team's discretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.